CLINICAL TRIAL: NCT02833376
Title: Alcohol 70% Versus Chlorhexidine 0.5% in the Spinal Anesthesia Skin Antissepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Luiz Carlos Tostes, MD, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MPLCT
Record Dates: First submitted 2016-07-05; First posted 2016-07-14 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2016-07

CONDITIONS: Anesthesia, Spinal; Anesthesia, Epidural; Antisepsis
Keywords: microbiota; ethanol; chlorhexidine
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alcohol group (Experimental): Patients allocated to this group will receive skin antisepsis with alcohol 70% prior spinal anesthesia
  Interventions: Other: alcohol antisepsis
- Chlorhexidine group (Experimental): Patients allocated to this group will receive skin antisepsis with alcoholic solution of chlorhexidine 0.5% prior spinal anesthesia
  Interventions: Other: chlorhexidine antisepsis

INTERVENTIONS:
Other: alcohol antisepsis
  Arms: Alcohol group
Other: chlorhexidine antisepsis
  Arms: Chlorhexidine group

SUMMARY:
Context: The neuraxial blocks, spinal anesthesia and epidural anesthesia are among the most frequently performed procedures worldwide, and despite the advancements of medical equipment, remain dependent on experience and practice of the anesthesiologists. Although antisepsis takes part of the daily routine, there are still no solid scientific evidence of the most appropriate antiseptic for these procedures.

Objective: To compare the 70% alcohol and 0.5% chlorhexidine alcohol solution in skin antisepsis for the neuraxial blocks.

Methods: This is a clinical trial, a prospective, randomized study. There will be selected, consecutively, 70 patients candidates for neuraxial blocks. Patients will be randomly assigned to group A (n = 35), in which the antisepsis will be performed with alcohol 70%, and to group B (n = 35), in which the antiseptic will be performed with the 0.5% chlorhexidine in alcoholic solution. Samples will be collected with swabs in an area of 25 cm² for bacterial cultures three times: in pre-antisepsis moments, in the second minute after antisepsis, and immediately after the puncture. The number of colonies forming units per square centimeter (CFU / cm²) will be counted. The data will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years of age , without restriction as to sex, ethnicity, education or social class;
* Patients who are undergoing neuraxial blockade by indicating the anesthesiologist responsible for the procedure

Exclusion Criteria:

* comorbidities or conditions which constitute a contraindication for the neuroaxial block ;
* Body mass index (BMI ) greater than 30 kg / m2;
* Ongoing infection;
* Use of antibiotics in the last seven days;
* Skin lesions at the puncture site ;
* Refusal to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Skin colonization before and after antisepsis, Will be counted number of colonies forming units per square centimeter (CFU/cm²) | Before antisepsis
  The material will be collected in a pre determined field of 25 cm², with a swab, and the maximum seeding in 8 hours, 48 hours after will be counted the number of colonies forming units per square centimeter (CFU/cm²)
Skin colonization before and after antisepsis, Will be counted number of colonies forming units per square centimeter (CFU/cm²) | 2 minutes after antisepsis
  The material will be collected in a pre determined field of 25 cm², with a swab, and the maximum seeding in 8 hours, 48 hours after will be counted the number of colonies forming units per square centimeter (CFU/cm²)
Skin colonization before and after antisepsis, Will be counted number of colonies forming units per square centimeter (CFU/cm²) | After the Puncture and at most 40 minutes
  The material will be collected in a pre determined field of 25 cm², with a swab, and the maximum seeding in 8 hours, 48 hours after will be counted the number of colonies forming units per square centimeter (CFU/cm²)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela F Veiga, MD, PhD, Study Chair — Universidade do Vale do Sapucai; Ana Beatriz A Loyola, PhD, Study Director — Universidade do Vale do Sapucai
Locations (1):
- Hospital e Maternidade Santa Paula, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tostes LCS, Loyola ABAT, Fraga AO, Gazzi LA, Paiva LF, Juliano Y, Veiga DF. Alcohol (70%) versus alcoholic chlorhexidine solution (0.5%) in skin antisepsis for neuraxial blocks: a randomized clinical trial. Rev Col Bras Cir. 2021 Jan 13;48:e20202633. doi: 10.1590/0100-6991e-20202633. eCollection 2021. PMID 33470369